CLINICAL TRIAL: NCT01362387
Title: R U OK? The Acceptability and Feasibility of New Communication Technologies for Follow-up After Medical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: British Pregnancy Advisory Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1.4.3
Record Dates: First submitted 2011-05-02; First posted 2011-05-30 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2011-05

CONDITIONS: Legally Induced Abortion, Complete, Without Mention of Complication
Keywords: Medical abortion; abortion follow-up

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (No Intervention): Women assigned to Group 1 will receive the standard post-abortion follow-up currently used at bpas and will be undertaken as usual by staff at the treating clinic
- Group 2 (Experimental): Follow-up after medical abortion using a standard text message, online or telephone questionnaire and a low sensitivity urine pregnancy test.
  Interventions: Other: Alternative follow-up protocol

INTERVENTIONS:
Other: Alternative follow-up protocol — Women (n=1000) will be allocated by chance to one of two groups: alternative follow-up using a standard text message, online or telephone questionnaire and a low sensitivity urine pregnancy test, or standard follow-up which consists of an in person visit with an ultrasound or a telephone call and high sensitivity pregnancy test.
  Arms: Group 2

SUMMARY:
Purpose: This randomised trial will compare outcomes and acceptability of an alternative medical abortion follow-up protocol using standardised text messaging, on-line questionnaire, or a phone interview and a low sensitivity pregnancy test with the current standard of care which consists of either a clinic visit and ultrasound scan or a telephone call and high sensitivity pregnancy test.

Hypothesis: The use of "alternative" methods to assess outcomes after early medical abortion will achieve a higher rate of follow-up than women undergoing "standard" follow-up

Primary aim: To determine the follow-up rate after early medical abortion with an alternative protocol as compared to a standard follow-up protocol

Secondary aims:

* To assess complication rates and receipt of further treatment among women in the two study arms
* To ascertain women's preferences for mode of communication regarding their post-medical abortion status
* To determine provider opinions and preferences for different follow-up modalities

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older,
* eligible for an abortion under the terms of the Abortion Act (1967),
* requesting an early medical abortion,
* willing and able to comply with the study protocol and visit schedule,
* access to either a mobile phone, intranet or telephone and willing to have communication by one of these means to assess post-medical abortion status,
* willing to have call back messages left,
* willing and able to provide valid informed consent, and
* able to communicate in English.

Exclusion Criteria:

* prior participation in this research study, or
* current participation in another research study that, in the opinion of the investigator, would interfere with the conduct of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 999 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of women with complete clinical information on post-abortion status | 14 days
  The primary purpose of this trial is to compare the ability of the two systems to identify the number of women who require additional medical abortion-related care.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Bracken, PhD, Principal Investigator — Gynuity Health Projects
Locations (4):
- United Kingdom (4):
  - Birmingham Day Care Unit, Birmingham
  - Chester Day Care Unit, Chester
  - London Central Day Care Unit, London
  - Luton Day Care Unit, Luton